CLINICAL TRIAL: NCT05818046
Title: Analysis of Arterial Waveforms and Oxygen Pressure During Supervised Exercise for Peripheral Artery Disease
Acronym: WAVESUPEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20-162
Record Dates: First submitted 2023-02-10; First posted 2023-04-18 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Supervised exercise therapy; arterial waveform; transcutaneous oxygen pressure
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Assignment (Experimental): intervention consiste to non-invasive arterial assessment by doppler (arterial waveform) and external oxygen probe (Transcutaneous oxygen pressure) at 3,6 and 9 weeks of supervised exercise therapy
  Interventions: Diagnostic Test: transcutaneous oxygen pressure; Procedure: Supervised Exercise therapy

INTERVENTIONS:
Diagnostic Test: transcutaneous oxygen pressure — External proxe fixed to the skin and ultrasound examination.
  Other Names: Doppler arterial waveform
Procedure: Supervised Exercise therapy — Supervised exercise therapy consists of three exercise sessions per week for 3 months, combining treadmill walking, lower limb muscle strengthening and stretching exercises. It is considered highly effective for people with leg pain related to peripheral arterial disease and has shown statistically significant improvements in maximum walking distance and quality of life parameters.

SUMMARY:
The goal of this observational study is to assess the evolution of oxygen pressure and arterial waveform during supervised exercise therapy in patients with peripheral arterial disease. The main questions it aims to answer are:

* can a significant increase in oxygen pressure be observed at 3 weeks?
* can a significant increase of oxygen pressure or arterial waveform be observed at 3, 6 or 9 weeks?

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a frequent pathology that affects more than 200 million people worldwide, more than 800,000 in France, and is mainly of atheromatous origin. The prevalence of this disease in France is estimated at 11% in people over 40 years of age, with an annual additional cost of €11,000 per patient. Supervised exercise therapy (SET) is the first-line treatment for intermittent claudication PAD for at least 3 months, although 15-20% of patients will not benefit from this therapy. Ankle-Brachial Index, the main diagnostic and monitoring tool for PAD, is not altered during SET. Transcutaneous oximetry (TcPO2) has been used for many years in the diagnosis of chronic permanent ischaemia, in the choice of amputation level and more recently in the diagnosis of proximal PAD.

No studies have investigated the evolution and predictive value of exercise TcPO2 in this context of SET. The assessment of arterial Doppler waveform using an objective classification has also never been performed in the specific context of SET. .

The goal of this observational study is to assess the evolution of oxygen pressure and arterial waveform during supervised exercise therapy in patients with peripheral arterial disease. The main questions it aims to answer are:

* can a significant increase in oxygen pressure be observed at 3 weeks?
* can a significant increase of oxygen pressure or arterial waveform be observed at 3, 6 or 9 weeks.

The perspective is to predict the effectiveness of SET in terms of maximum walking distance.

ELIGIBILITY:
Inclusion Criteria:

* PAD with intermittent claudication
* SET prescribed
* ABI < 0.9
* Beneficiary of French health care insurance

Exclusion Criteria:

* PAD with rest ischemia
* Chronic respiratory failure
* Acute decompensated disease
* Lower limb prosthesis
* Pregnant women and breastfeeding mothers
* Place of residence more than 100 km from Caen University Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Evolution of oximetry at 3 week from baseline | at 3 weeks
  To describe the evolution of oximetry during SET at 3 weeks from baseline (TcPO2 leg value)

SECONDARY OUTCOMES:
Evolution of doppler waveform at 3 week from baseline | at 3 weeks
  To describe the evolution of doppler waveform during SET at 3 weeks from baseline (SB hemodynamic classification)
Evolution of doppler waveform at 6 week from baseline | 6 weeks
  To describe the evolution of doppler waveform during SET at 6 weeks from baseline (SB hemodynamic classification)
Evolution of doppler waveform at 9 week from baseline | 9 weeks
  To describe the evolution of doppler waveform during SET at 9 weeks from baseline (SB hemodynamic classification)
Evolution of doppler waveform at 12 week from baseline | 12 weeks
  To describe the evolution of doppler waveform during SET at 12 weeks from baseline (SB hemodynamic classification)
Evolution of oximetry at 6 week from baseline | at 6 weeks
  To describe the evolution of oximetry during SET at 6 weeks from baseline (TcPO2 leg value)
Evolution of oximetry at 9 week from baseline | at 9 weeks
  To describe the evolution of oximetry during SET at 9 weeks from baseline (TcPO2 leg value)
Evolution of oximetry at 12 week from baseline | at 12 weeks
  To describe the evolution of oximetry during SET at 12 weeks from baseline (TcPO2 leg value)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] STRANDNESS DE Jr, BELL JW. AN EVALUATION OF THE HEMODYNAMIC RESPONSE OF THE CLAUDICATING EXTREMITY TO EXERCISE. Surg Gynecol Obstet. 1964 Dec;119:1237-42. No abstract available. PMID 14227748
- [Background] Gardner AW. Reliability of transcutaneous oximeter electrode heating power during exercise in patients with intermittent claudication. Angiology. 1997 Mar;48(3):229-35. doi: 10.1177/000331979704800305. PMID 9071198
- [Background] Spronk S, den Hoed PT, de Jonge LC, van Dijk LC, Pattynama PM. Value of the duplex waveform at the common femoral artery for diagnosing obstructive aortoiliac disease. J Vasc Surg. 2005 Aug;42(2):236-42; discussion 242. doi: 10.1016/j.jvs.2005.04.048. PMID 16102620
- [Background] Mahe G, Boulon C, Desormais I, Lacroix P, Bressollette L, Guilmot JL, Le Hello C, Sevestre MA, Pernod G, Constans J, Boissier C, Bura-Riviere A. Statement for Doppler waveforms analysis. Vasa. 2017 Aug;46(5):337-345. doi: 10.1024/0301-1526/a000638. Epub 2017 May 19. PMID 28521662
- [Background] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FG, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RA, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Mar 21;135(12):e726-e779. doi: 10.1161/CIR.0000000000000471. Epub 2016 Nov 13. PMID 27840333
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I; ESC Scientific Document Group. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS): Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteriesEndorsed by: the European Stroke Organization (ESO)The Task Force for the Diagnosis and Treatment of Peripheral Arterial Diseases of the European Society of Cardiology (ESC) and of the European Society for Vascular Surgery (ESVS). Eur Heart J. 2018 Mar 1;39(9):763-816. doi: 10.1093/eurheartj/ehx095. No abstract available. PMID 28886620